CLINICAL TRIAL: NCT00028340
Title: Characterization of High-Risk Breast Duct Epithelium by Cytology, Breast Duct Endoscopy, and cDNA Gene Expression Profile
Brief Title: High-Risk Breast Duct Epithelium
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020077; 02-C-0077; NCT00070460 (obsolete NCT alias)
Record Dates: First submitted 2001-12-21; First posted 2001-12-24 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Natural History
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Breast Cancer and High-Risk Patients: Pre- or postmenopausal women who have or have previously had invasive or noninvasive breast cancer of epithelial origin, or women without breast cancer but at an increased risk of breast cancer.
- 2/Normal Volunteers: Pre- or postmenopausal women who are not at an increased risk for breast cancer.

SUMMARY:
Background:

* Breast cancer is the most common malignancy in women, occurring in over 230,000 women annually in the United States.
* The vast majority of breast cancers originate in the single layer of epithelial cells that line the ductal/lobular system of the breast milk ducts. The premalignant changes which occur in the transformed epithelium are not well understood, however several cytologic or histologic changes have been identified which are associated with an increased risk for breast cancer, including ductal or lobular hyperplasia, hyperplasia with atypia, and lobular or ductal carcinoma in situ.
* The identification of cytological or histological abnormalities in breast epithelial cells is an important component of risk assessment.

Objective:

Primary objectives are:

* To determine the incidence and nature of cytologic changes in ductal epithelial cells from the high-risk breast, in specimens collected by breast ductal lavage, and to determine if these cytologic findings are different from those of female normal volunteers not at increased risk for breast cancer.
* To characterize by breast duct endoscopy, high risk breast ductal epithelium and architecture, and correlate these findings with the cytologic findings referenced in above bullet.
* To determine what is the global gene expression pattern of high risk breast epithelial cells from the high risk breast, and does this differ from that of breast epithelial cells from female normal volunteersnot at increased risk for breast cancer. The gene expression profile will be determined by cDNA microarray and validated by RT-PCR.

Eligibility:

Eligibility for high risk individuals will include:

* Women with a unilateral invasive or noninvasive (DCIS) breast cancer of epithelial origin.
* Women without breast cancer, but with a Gail Index greater than 1.67 percent, or a cumulative lifetime risk greater than or equal to double the age- and race-matched general population risk.
* Women known to be BRCA1/2 or other hereditary genes mutation carriers.
* Women with cytologic or histologic evidence of ductal hyperplasia, atypical ductal hyperplasia, or lobular carcinoma in situ.
* Women may be either premenopausal or postmenopausal. Postmenopausal is defined by the absence of menstrual periods for at least 12 months.
* Postmenopausal women who have previously undergone a hysterectomy without oophorectomy must have a serum FSH level of > 40 IU/ml, and a serum estradiol level of less than40 pg/ml to document postmenopausal status.

Eligibility for normal volunteers will include:

* Women who are premenopausal or postmenopausal with a Gail model risk index less than 1.67 percent, and without a cumulative lifetime risk greater than or equal to double the age- and racematched general population risk.
* Women who have previously undergone a hysterectomy without oophorectomy must have a serum FSH level of >40 IU/ml, and a serum estradiol level of less than 40 pg/ml to document postmenopausal status.
* Both breasts must be free of any suspicious areas by physical examination and, for women over 30 years of age by mammogram. There must be no history of atypical hyperplasia, invasive or in situ carcinoma.

Both groups must have acceptable white blood cell and platelet counts.

Design:

Breast ductal epithelial cells will be collected by breast ductal lavage from (a) the breast in women at increased risk for breast cancer, and (b) the breast of female normal volunteers who are not at increased risk for breast cancer.

Ductal epithelial cell specimens will be analyzed cytologically for the presence of hyperplasia, atypia, or in situ changes.

Breast duct endoscopy will be performed in breast cancer patients and in normal volunteers with cytologic atypia on ductal lavage to determine ductal architectural changes associated with increased risk for breast cancer, and to provide correlation with cytologic atypia.

The gene expression profile of normal and high-risk ductal epithelial cells will be studied by cDNA-microarray to determine changes in gene expression associated with increased risk for breast cancer.

Additional molecular profiling experiments which will be performed as lavage cells are available include DNA whole exome sequencing, Comparative Genomic Hybridization (CGH), proteomic tissue lysate arrays, and identification of mammary stem cells.

A total of 104 high-risk subjects and 110 normal volunteers will be studied, divided approximately evenly between premenopausal and postmenopausal women....

DETAILED DESCRIPTION:
Background:

Breast cancer is the most common malignancy in women, occurring in over 230,000 women annually in the United States.

The vast majority of breast cancers originate in the single layer of epithelial cells that line the ductal/lobular system of the breast milk ducts. The premalignant changes which occur in the transformed epithelium are not well understood: however, several cytologic or histologic changes have been identified which are associated with an increased risk for breast cancer, including ductal or lobular hyperplasia, hyperplasia with atypia, and lobular or ductal carcinoma in situ.

The identification of cytological or histological abnormalities in breast epithelial cells is an important component of risk assessment.

Objective:

Primary objectives:

To determine the incidence and nature of cytologic changes in ductal epithelial cells from the high-risk breast, in specimens collected by breast ductal lavage, and to determine if these cytologic findings are different from those of female normal volunteers not at increased risk for breast cancer.

To characterize by breast duct endoscopy high-risk breast ductal epithelium and architecture, and correlate these findings with the cytologic findings referenced in above bullet.

To determine what is the global gene expression pattern of high-risk breast epithelial cells from the high-risk breast, and does this differ from that of breast epithelial cells from female normal volunteers not at increased risk for breast cancer. The gene expression profile will be determined by cDNA microarray and validated by RT-PCR.

Eligibility:

Eligibility for high-risk individuals will include:

Women with a unilateral invasive or noninvasive (DCIS) breast cancer of epithelial origin.

Women without breast cancer, but with a Gail Index > 1.67 percent, or a cumulative lifetime risk greater than or equal to double the age- and race-matched general population risk.

Women known to be BRCA1/2 or other hereditary genes mutation carriers.

Women with cytologic or histologic evidence of ductal hyperplasia, atypical ductal hyperplasia, or lobular carcinoma in situ.

Women may be either premenopausal or postmenopausal. Postmenopausal is defined by the absence of menstrual periods for at least 12 months.

Postmenopausal women who have previously undergone a hysterectomy without oophorectomy must have a serum FSH level of > 40 IU/mL, and a serum estradiol level of < 40 pg/mL to document postmenopausal status.

Eligibility for normal volunteers will include:

Women who are premenopausal or postmenopausal with a Gail model risk index < 1.67 percent, and without a cumulative lifetime risk greater than or equal to double the age- and race-matched general population risk.

Women who have previously undergone a hysterectomy without oophorectomy must have a serum FSH level of > 40 IU/mL, and a serum estradiol level of < 40 pg/mL to document postmenopausal status.

Both breasts must be free of any suspicious areas by physical examination and, for women over 30 years of age, by mammogram. There must be no history of atypical hyperplasia, invasive, or in situ carcinoma.

Both groups must have acceptable white blood cell and platelet counts.

Design:

Breast ductal epithelial cells will be collected by breast ductal lavage from (a) the breast in women at increased risk for breast cancer, and (b) the breast of female normal volunteers who are not at increased risk for breast cancer.

Ductal epithelial cell specimens will be analyzed cytologically for the presence of hyperplasia, atypia, or in situ changes.

Breast duct endoscopy will be performed in breast cancer patients and in normal volunteers with cytologic atypia on ductal lavage to determine ductal architectural changes associated with increased risk for breast cancer, and to provide correlation with cytologic atypia.

The gene expression profile of normal and high-risk ductal epithelial cells will be studied by cDNA microarray to determine changes in gene expression associated with increased risk for breast cancer.

Additional molecular profiling experiments which will be performed as lavage cells are available include DNA whole exome sequencing, comparative genomic hybridization (CGH), proteomic tissue lysate arrays, and identification of mammary stem cells.

A total of 104 high-risk subjects and 110 normal volunteers will be studied, divided approximately evenly between premenopausal and postmenopausal women.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Breast Cancer and High-Risk Patients:

* Age greater than or equal to 18 years and less than or equal to 74 years.

  * Women with a unilateral invasive or noninvasive (DCIS) breast cancer of epithelial origin.
  * Women without breast cancer, but with a Gail Index greater than 1.67 percent, or a cumulative lifetime risk greater than or equal to double the age- and race-matched general population risk.
  * Women known to be BRCA1/2 or other hereditary genes mutation carriers.
  * Women with cytologic or histologic evidence of ductal hyperplasia, atypical ductal hyperplasia, or LCISl
  * Women may be either premenopausal or postmenopausal. Postmenopausal is defined by the absence of menstrual periods for at least 12 months.
  * Postmenopausal women who have previously undergone a hysterectomy without oophorectomy must have a serum FSH level of greater than 40 IU/ml, and a serum estradiol level of less than 40 pg/ml to document postmenopausal status.
  * Breast cancer may be invasive or noninvasive, and in the past or the present.
  * The contralateral breast of women with breast cancer, or the normal breast of high-risk subjects, must be free of any suspicious areas by physical examination and mammogram, and without a history of invasive ductal or in situ ductal carcinoma. History of atypia or LCIS on a previous biopsy is acceptable.
  * Women who are from a family with heritable breast cancer with a known deleterious BRCA1/2 or other hereditary genes mutation, who themselves have been tested and to not carry this mutation. These women are not at increased risk for breast cancer due to the familial mutation and are eligible to participate as normal volunteers.
  * WBC greater than 2,500.
  * Platelets greater than 50,000.
* Inclusion Criteria for Normal Volunteers:
* Age greater than or equal to 18 years and less than or equal to 74 years.

  * Women who are premenopausal or postmenopausal with a Gail model risk index less than 1.67 percent, and without a cumulative lifetime risk greater than or equal to double the age- and race-matched general population risk.
  * Women who have previously undergone a hysterectomy without oophorectomy must have a serum FSH level of greater than 40 IU/ml, and a serum estradiol level of less than 40 pg/ml to document postmenopausal status.
  * Both breasts must be free of any suspicious areas by physical examination and, for women over 30 years of age by mammogram. There must be no history of atypical hyperplasia, invasive or in situ carcinoma.
  * WBC greater than 2,500.
  * Platelets greater than 50,000.

EXCLUSION CRITERIA:

* Exclusion Criteria for Breast Cancer Patients:

  * Contralateral breast prosthesis
  * Pregnancy
  * History of radiation therapy to the contralateral breast
  * Lactating breasts
  * Chemotherapy within the past 1 month
  * Current antiestrogen therapy
  * Current hormonal replacement therapy or oral contraceptives
  * Concurrent infection
  * Previous contralateral major duct excision
* Exclusion Criteria for High-Risk Paitents:

  * Bilateral breast prosthesis
  * Pregnancy
  * Lactating breasts
  * Current antiestrogen therapy
  * Current hormonal replacement therapy or oral contraceptives
  * Concurrent infection
  * Previous bilateral major duct excision
  * History of therapeutic mediastinal radiation
* Exclusion Criteria for Normal Volunteers:

  * Bilateral breast prosthesis
  * Pregnancy
  * Lactating breasts
  * Current antiestrogen therapy
  * Current hormonal replacement therapy or oral contraceptives
  * Concurrent infection
  * Previous bilateral major duct excision
  * History of therapeutic mediastinal radiation

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre- or postmenopausal women who have or have previously had invasive or noninvasive breast cancer of epithelial origin, or women without breast cancer but at an increased risk of breast cancer. Pre- or postmenopausal women who are not at an increased risk for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2003-02-20 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Determine the incidence and nature of cytologic changes in ductal epithelial cells from the high-risk breast. | 25 years
  Using specimens collected by breast ductal lavage, and determine if these cytologic findings are different from those of normal women not at increased risk for breast cancer.
Determine the global gene expression pattern of high-risk breast epithelial cells from the high-risk breast. | 25 years
  Determine if gene expression pattern differs from that of breast epithelial cells from female normal volunteers not at increased risk for breast cancer. Gene expression profile will be determined by cDNA microarray and validated by RT-PCR.
Characterize high-risk breast ductal epithelium and architecture. | 25 years
  Characterize by breast duct endoscopy, and correlate these findings with the cytologic findings.

SECONDARY OUTCOMES:
Examine ductal epithelial cell preparations for the presence of mammary stem cells. | 25 years
  From both women at high risk and from women not at high risk for breast cancer.
Determine the pattern of protein expression for selected proteins in the high-risk epithelial cells. | 25 years
  Using proteomics tissue lysate arrays.
Determine the gross genomic alterations present in high-risk breast epithelial cells. | 25 years
  Using comparative genomic hybridization.
Determine the DNA mutational pattern of breast epithelium from women at high risk for breast cancer. | 25 years
  Using DNA whole exome sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: David N Danforth, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.@@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.@@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Fisher B, Costantino J, Redmond C, Fisher E, Margolese R, Dimitrov N, Wolmark N, Wickerham DL, Deutsch M, Ore L, et al. Lumpectomy compared with lumpectomy and radiation therapy for the treatment of intraductal breast cancer. N Engl J Med. 1993 Jun 3;328(22):1581-6. doi: 10.1056/NEJM199306033282201. PMID 8292119
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] Fisher B, Dignam J, Wolmark N, Wickerham DL, Fisher ER, Mamounas E, Smith R, Begovic M, Dimitrov NV, Margolese RG, Kardinal CG, Kavanah MT, Fehrenbacher L, Oishi RH. Tamoxifen in treatment of intraductal breast cancer: National Surgical Adjuvant Breast and Bowel Project B-24 randomised controlled trial. Lancet. 1999 Jun 12;353(9169):1993-2000. doi: 10.1016/S0140-6736(99)05036-9. PMID 10376613
- [Derived] Danforth DN, Filie AC, Warner AC, Wright GW, Sun Z, Ried T, McGowan CT, Prindiville SA. Characteristics of Breast Ducts in Normal-Risk and High-risk Women and Their Relationship to Ductal Cytologic Atypia. Cancer Prev Res (Phila). 2020 Dec;13(12):1027-1036. doi: 10.1158/1940-6207.CAPR-19-0305. Epub 2020 Aug 4. PMID 32753377
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0077.html